CLINICAL TRIAL: NCT07001163
Title: Assessment of the Role of Probiotics in Prevention of Ventilator-Associated Pneumonia in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lamiaa Khaled Zidan (Other)
Responsible Party: Sponsor-Investigator, Lamiaa Khaled Zidan, Lecturer, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Probiotics in neonatal VAP
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Ventilator Acquired Pneumonia
Keywords: VAP, NICU
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Active Comparator): 40 ventilated neonates who received commercially available probiotics
  Interventions: Dietary Supplement: Probiotic
- Non-probiotic group (No Intervention): 40 ventilated neonates who only received the standard of care treatment

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic sachets contained 1× 109 colony-forming unit of Bifidobacterium Animalis subsp.lactis BB-12), were given via orogastric tube twice daily.
  Arms: Probiotic group

SUMMARY:
Evaluate the preventive value of probiotics on VAP among ventilated neonates.

DETAILED DESCRIPTION:
MV is a critical component of neonatal intensive care, providing essential respiratory support for neonates with severe respiratory distress. However, its use is associated with an increased risk of VAP, a serious nosocomial lung infection. VAP is defined as a pneumonia diagnosed in patients undergoing MV for at least 48 hours and is recognized as the second most common nosocomial infection in neonatal and pediatric intensive care units. Its incidence ranges from 1 to 63 episodes per 1,000 ventilation days, with variability influenced by the socioeconomic and healthcare development of different regions.Given the complex pathophysiology of VAP, numerous prevention strategies have been proposed for NICUs.Among these strategies, probiotics have emerged.

ELIGIBILITY:
Inclusion Criteria:

* All term neonates who required mechanical ventilation with ETT for more than 48 hours.

Exclusion Criteria:

1. Early-onset neonatal sepsis
2. Pre-existing pneumonia
3. A patient who was unfit for enteral intake.
4. Prematurity <37 gestational weeks.
5. Surgical causes of mechanical ventilation
6. Multiple congenital anomalies and suspected chromosomal anomalies.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
VAP incidence rate | one year
  Evaluation of the role of probiotics in the Prevention of neonatal VAP and examining their impact on the incidence of VAP at those neonates.

SECONDARY OUTCOMES:
GIT manifestations | one year
  Evaluation of the effect of probiotics in critically ventilated neonates on the incidence of GIT manifestations as Feeding intolerance, Vomiting, Constipation, or diarrhea.
Duration of MV and NICU stay | one year
  Assessment of the impact of probiotic supplementation on critically ventilated neonates in terms of mechanical ventilation duration and NICU length of stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Tanta University, Tanta, Q2x2+cp Tanta 2, Egypt,, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bondarev DJ, Ryan RM, Mukherjee D. The spectrum of pneumonia among intubated neonates in the neonatal intensive care unit. J Perinatol. 2024 Sep;44(9):1235-1243. doi: 10.1038/s41372-024-01973-9. Epub 2024 May 2. PMID 38698211
- [Background] Iqbal F, Siva N, Kolibylu Raghupathy M, Edward S Lewis L, Barche A, Purkayastha J, S Nayak B. Probiotic effect in preterm neonates with sepsis - A systematic review protocol. F1000Res. 2024 Jul 5;11:913. doi: 10.12688/f1000research.122226.3. eCollection 2022. PMID 39114384
- [Background] Rangelova V, Kevorkyan A, Raycheva R, Krasteva M. Ventilator-Associated Pneumonia in the Neonatal Intensive Care Unit-Incidence and Strategies for Prevention. Diagnostics (Basel). 2024 Jan 23;14(3):240. doi: 10.3390/diagnostics14030240. PMID 38337756
- [Derived] Khodair HA, Elmahdy HS, Zidan LK, Elashry SM, Elmashad AEM. Assessment of the role of probiotics in prevention of ventilator-associated pneumonia in neonates. Eur J Pediatr. 2025 Sep 4;184(9):597. doi: 10.1007/s00431-025-06380-6. PMID 40906025